CLINICAL TRIAL: NCT04194580
Title: Effectiveness of a Physical Activity Intervention on the Overweight and Obesity of Chilean Schoolchildren
Brief Title: Physical Activiy Intervention Programm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autónoma de Chile (Other)
Responsible Party: Principal Investigator, Andrés Godoy Cumillaf, Profesor, Universidad Autónoma de Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAChile
Record Dates: First submitted 2019-12-03; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Physical Activity; Fitness; Overweight and Obesity
MeSH Terms: conditions — Motor Activity; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity (Experimental): In the program we will perform a recreational physical activity intervention during one year that include standardized recreative and non competitive activities conducted by sports instructors
  Interventions: Behavioral: Phisical activity intervention
- Physical activity control (No Intervention): This group will not participate in the intervention

INTERVENTIONS:
Behavioral: Phisical activity intervention — The prevalence of overweight in chilean children in the among the highest in the world and increasing quickly. The investigators recently evaluated an after-school program of recreational physical activity to control overweight, obesity and other cardiovascular risk factors in primary school children Temuco. This program reduced adiposity and increased the fitness.
  Arms: Physical activity

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a recreational physical activity intervention for reducing the prevalence of overweight/obesity and other cardiovascular risk factors

DETAILED DESCRIPTION:
A greater intensity of the intervention, and a longer weekly duration that extends until the weekend, could improve the efficiency in obesity.

ELIGIBILITY:
Inclusion Criteria:

* The parents of the children will be informed about the objectives and methods of the study, and will give their written consent to the participation of the children. Similarly, the study will introduce children from classroom to class and their oral consent will be obtained

Exclusion Criteria:

* Participating children will be free from serious learning difficulties, or physical or mental disorders, that could prevent participation in scheduled physical activities.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Aerobic Capacity | 1 year
  By using 20-m shuttle run test, which is validated to measure maximal aerobic capacity in children from 4 years.
Muscle Strength | 1 year
  By using standing long jump test
Flexibility | 1 year
  By using the sit and reach test
Speed-agility | 1 year
  By using 4x10 meters shuttle run test

SECONDARY OUTCOMES:
Health-related quality of life | 1 year
  By using the instrument for assessing Health-Related Quality of Life for children and adolescents aged 4-17 years (KINDL), in its version validated in Spanish. The KINDLR questionnaire consists of 24 Likert-scaled items associated with six dimensions: physical well-being, emotional well-being, self-esteem, family, friends and everyday functioning (school or nursery school/kindergarten). The sub-scales of these six dimensions can be combined to produce a total score. the score ranges from 0 to 100. Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: José Bruneau, PhD, Study Director — Universidad Autónoma de Chile
Locations (1):
- Laboratorio Fisiología del Ejercicio, Temuco, La Araucanía, Chile

REFERENCES:
- [Derived] Godoy-Cumillaf A, Fuentes-Merino P, Giakoni-Ramirez F, Duclos-Bastias D, Merellano-Navarro E. Effectiveness of a physical activity intervention on the overweight and obesity of Chilean schoolchildren. Medicine (Baltimore). 2022 Sep 30;101(39):e30908. doi: 10.1097/MD.0000000000030908. PMID 36181063